CLINICAL TRIAL: NCT02937454
Title: A Randomised, Double-Blind Placebo Controlled Trial Comparing the Effect of Intravenous Ferric Carboxymaltose on Hospitalisations and Mortality in Iron Deficient Patients Admitted for Acute Heart Failure (Affirm-AHF)
Brief Title: Study to Compare Ferric Carboxymaltose With Placebo in Patients With Acute Heart Failure and Iron Deficiency
Acronym: Affirm-AHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vifor (International) Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other); Cytel Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FER-CARS-06; 2016-001467-36 (EudraCT Number)
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Iron Deficiency; Heart Failure
Keywords: Acute Heart Failure; Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies; Heart Failure | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ferric carboxymaltose (Active Comparator): The first dose of study treatment will be administered for all randomised subjects while the patient is still hospitalised for the Index hospitalisation. The subsequent administrations of study treatment will be done as part of the outpatient clinic visits.
  Interventions: Drug: ferric carboxymaltose
- normal saline 0.9% (Placebo Comparator): The first dose of study treatment will be administered for all randomised subjects on the same day as randomisation.
  Interventions: Other: Normal saline 0.9%

INTERVENTIONS:
Drug: ferric carboxymaltose — FCM will be administered as an undiluted bolus injection. The study treatment dose (mL) to be administered will be determined by the patient's body weight and haemoglobin (Hb) value at the respective visits where study treatment will be administered
  Other Names: Injectafer; Ferinject; Renegy; Iroprem
  Arms: ferric carboxymaltose
Other: Normal saline 0.9% — Normal saline will be administered as a bolus injection.
  Arms: normal saline 0.9%

SUMMARY:
Study to Compare Ferric Carboxymaltose With Placebo in Patients With Acute Heart Failure and Iron Deficiency (Affirm-AHF)

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled Trial (RCT). The 52 weeks observation period following randomisation is considered appropriate to investigate the primary endpoint of recurrent HF hospitalisations and CV death. To evaluate the effect of intravenous ferric carboxymaltose (IV FCM) in iron deficient subjects with AHF, subjects will be enrolled during a hospital stay (Index hospitalisation) after the acute care treatment of the index event has been stabilised. All subjects will continue to receive their established standard therapy for HF and medical emergencies will be treated according to local routine.

ELIGIBILITY:
Inclusion Criteria:

1. Currently hospitalised for an episode of acute heart failure (AHF) where AHF was the primary reason for hospitalisation. All of the following (i.e., items a to d) must apply:

   1. Upon admission for the AHF episode, persistent dyspnoea at rest in a recumbent sitting position (30-45°) or with minimal exertion
   2. Upon or during the AHF admission, at least 2 of the following clinical findings were present: i. Congestion on chest X-ray ii. Rales on chest auscultation iii. Oedema ≥1+ on a 0-3+ scale, indicating indentation of skin with mild digital pressure that requires 10 or more seconds to resolve in any dependent area including extremities or sacral region iv. Elevated jugular venous pressure (≥8 cm H2O)
   3. Natriuretic peptide levels, measured ≤72 hours of the AHF admission must have been: i. Brain natriuretic peptide (BNP) ≥400 pg/mL or N-terminal-pro-brain natriuretic peptide (NT-proBNP) ≥1,600 pg/mL or ii. BNP ≥600 pg/mL or NT-proBNP ≥2,400 pg/mL for subjects presenting with atrial fibrillation when the blood sample was taken iii. For subjects treated with an angiotensin receptor neprilysin inhibitor (ARNI) in the previous 4 weeks prior to randomisation only NT-proBNP values should be considered
   4. AHF episode treated with minimally 40 mg of IV furosemide (or equivalent IV loop diuretic defined as 20 mg of torasemide or 1 mg of bumetanide)
2. Subject is iron deficient defined as serum ferritin <100 ng/mL or 100 ng/mL ≤ serum ferritin ≤299 ng/mL if TSAT <20%.
3. Left ventricular ejection fraction <50% (assessed and documented within 12 months prior to randomisation).
4. Male or female aged ≥18 years old.
5. Subject (or legally acceptable representative)* has provided the appropriate written informed consent. Subject must provide written informed consent before any study-specific procedures are performed.

Exclusion Criteria:

1. Dyspnoea due to non-cardiac causes such as acute or chronic respiratory disorders or infections (i.e., severe chronic obstructive pulmonary disease, acute bronchitis, pneumonia, primary pulmonary hypertension).
2. Temperature >38°C (oral or equivalent), active infective endocarditis, sepsis, systemic inflammatory response syndrome, or any other active infection requiring anti-microbial treatment at any time during an Index hospitalisation. (Note that it does NOT include short-term prophylactic administration of antibiotics or short-term temperature elevation at admission which is no longer present at the time point of discharge/randomisation).
3. Documented restricted amyloid myocardiopathy, or acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy. (Note that it does NOT include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).
4. Clinical evidence of acute coronary syndrome, transient ischemic attack or stroke, within the last 30 days prior randomisation.
5. Severe valvular or left ventricular outflow obstruction disease needing intervention.
6. Coronary-artery bypass graft, cardiac resynchronisation therapy device implantation, percutaneous intervention (e.g., cardiac, cerebrovascular, aortic, diagnostic catheters are allowed) or major surgery that led to significant blood loss, including thoracic and cardiac surgery, within the last 3 months prior to randomisation.
7. Subject has a body weight <35 kg at randomisation.
8. Subject at an immediate need of transfusion or with a Hb <8 g/dL* or with a Hb >15 g/dL.
9. Subjects on treatment for Vitamin B12 and/or serum folate deficiency. Note: Use of Vitamin B12 and folic acid as supplement therapy (not for deficiency treatment) is permitted.
10. Subject with a known anaemia not attributed to ID (e.g., other microcytic anaemia) or with an evidence of iron overload (e.g., haemochromatosis) or disturbances in the utilisation of iron.
11. Subject has known hypersensitivity to any of the study products to be administered or known serious hypersensitivity to other parenteral iron products.
12. Subject with known severe allergies including drug allergies, history of severe asthma, eczema or other atopic allergy and in subjects with immune or inflammatory conditions (e.g., systemic lupus erythematosus, rheumatoid arthritis).
13. History of erythropoietin stimulating agent, IV iron therapy, and/or blood transfusion in previous 3 months prior to randomisation.
14. Oral iron therapy at doses >100 mg/day in previous 4 weeks prior to randomisation. Note: Ongoing use of multivitamins containing iron <75 mg/day are permitted.
15. Currently receiving systemic chemotherapy and/or radiotherapy.
16. Renal dialysis (previous, current or planned within the next 6 months).
17. Subject has known active malignancy of any organ system, i.e., clinical evidence of current malignancy or not in stable remission for at least 3 years since completion of last treatment with exception of non-invasive basal cell carcinoma, squamous cell carcinoma of the skin or cervical intra-epithelial neoplasia.
18. Terminal illness other than HF with expected survival <12 months.
19. Chronic liver disease (including active hepatitis) and/or alanine transaminase or aspartate transaminase above 3 times the upper limit of the normal range.
20. Subjects with known hepatitis B surface antigen positivity and/or hepatitis C virus ribonucleic acid positivity.
21. Subject previously randomised into this study. Note: Subjects may be rescreened but when rescreened, all tests must fall inside the maximum specified screening windows for each criterion.
22. Subject is currently enrolled in or has completed any other investigational device or drug study <30 days prior to screening, or is receiving other investigational agent(s).
23. Subject is pregnant (e.g., positive human chorionic gonadotropin test) or breast feeding.
24. If of childbearing potential, subject is not using adequate contraceptive precautions. Subject must agree to use adequate contraception during the study and for 1 month after the last dose of study treatment. A highly effective method of birth control must be used.
25. Subject has a history of drug or alcohol abuse within 2 years prior to screening.
26. Subject has a significant medical condition(s), anticipated need for major surgery during the study, or any other kind of disorder that may be associated with increased risk to the subject, or may interfere with study assessments, outcomes, or the ability to provide written informed consent or comply with study procedures, in the Investigator's opinion.

    * Following section in italics is applicable for The Netherlands, Spain and Singapore only (NL, ES and SG only): 'The lower threshold of Hb values is set to 10 g/dL.'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1132 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, MD, Principal Investigator — Medical University Clinical Military Hospital
Locations (16):
- Hospital Universitario Austral, Buenos Aires, Argentina
- InCor -Instituto do Coração HCFMUSP, São Paulo, Brazil
- Clinical Hospital Center Rijeka, Rijeka, Croatia
- Aleksandre Aladashvili Clinic LLC, Tbilisi, Georgia
- Israel (2):
  - The Baruch Pade Medical Center, Tiberias, Lower Galilee
  - Hadassah Ein Kerem University Medical Center, Jerusalem
- Spedali Civilia di Brescia, Brescia, Italy
- American University of Beirut Medical Center, Beirut, Lebanon
- Vasculair Onderzoek Centrum, Hoorn, Netherlands
- Clinical Military Hospital, Wroclaw, Poland
- Emergency Clinical Hospital, Bucharest, Romania
- National Heart Centre of Singapore Pte, Singapore, Singapore
- University of Murcia, Murcia, Spain
- Skane University Hospital, Malmo, Sweden
- The M.D. Strazhesko Institute of Cardiology, Kyiv, Ukraine
- Kings College Hospital NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosano G, Ponikowski P, Vitale C, Anker SD, Butler J, Fabien V, Filippatos G, Kirwan BA, Macdougall IC, Metra M, Ruschitzka F, Kumpeson V, Goehring UM, van der Meer P, Jankowska EA; AFFIRM-AHF investigators. Intravenous ferric carboxymaltose for iron repletion following acute heart failure in patients with and without diabetes: a subgroup analysis of the randomized AFFIRM-AHF trial. Cardiovasc Diabetol. 2023 Aug 17;22(1):215. doi: 10.1186/s12933-023-01943-z. PMID 37592272
- [Derived] Macdougall IC, Ponikowski P, Stack AG, Wheeler DC, Anker SD, Butler J, Filippatos G, Gohring UM, Kirwan BA, Kumpeson V, Metra M, Rosano G, Ruschitzka F, van der Meer P, Wachter S, Jankowska EA. Ferric Carboxymaltose in Iron-Deficient Patients with Hospitalized Heart Failure and Reduced Kidney Function. Clin J Am Soc Nephrol. 2023 Sep 1;18(9):1124-1134. doi: 10.2215/CJN.0000000000000223. Epub 2023 Jun 29. PMID 37382961
- [Derived] Filippatos G, Ponikowski P, Farmakis D, Anker SD, Butler J, Fabien V, Kirwan BA, Macdougall IC, Metra M, Rosano G, Ruschitzka F, van der Meer P, Wachter S, Jankowska EA; AFFIRM-AHF Investigators. Association Between Hemoglobin Levels and Efficacy of Intravenous Ferric Carboxymaltose in Patients With Acute Heart Failure and Iron Deficiency: An AFFIRM-AHF Subgroup Analysis. Circulation. 2023 May 30;147(22):1640-1653. doi: 10.1161/CIRCULATIONAHA.122.060757. Epub 2023 Apr 13. PMID 37051919
- [Derived] Ponikowski P, Kirwan BA, Anker SD, McDonagh T, Dorobantu M, Drozdz J, Fabien V, Filippatos G, Gohring UM, Keren A, Khintibidze I, Kragten H, Martinez FA, Metra M, Milicic D, Nicolau JC, Ohlsson M, Parkhomenko A, Pascual-Figal DA, Ruschitzka F, Sim D, Skouri H, van der Meer P, Lewis BS, Comin-Colet J, von Haehling S, Cohen-Solal A, Danchin N, Doehner W, Dargie HJ, Motro M, Butler J, Friede T, Jensen KH, Pocock S, Jankowska EA; AFFIRM-AHF investigators. Ferric carboxymaltose for iron deficiency at discharge after acute heart failure: a multicentre, double-blind, randomised, controlled trial. Lancet. 2020 Dec 12;396(10266):1895-1904. doi: 10.1016/S0140-6736(20)32339-4. Epub 2020 Nov 13. PMID 33197395
- [Derived] Ponikowski P, Kirwan BA, Anker SD, Dorobantu M, Drozdz J, Fabien V, Filippatos G, Haboubi T, Keren A, Khintibidze I, Kragten H, Martinez FA, McDonagh T, Metra M, Milicic D, Nicolau JC, Ohlsson M, Parhomenko A, Pascual-Figal DA, Ruschitzka F, Sim D, Skouri H, van der Meer P, Jankowska EA. Rationale and design of the AFFIRM-AHF trial: a randomised, double-blind, placebo-controlled trial comparing the effect of intravenous ferric carboxymaltose on hospitalisations and mortality in iron-deficient patients admitted for acute heart failure. Eur J Heart Fail. 2019 Dec;21(12):1651-1658. doi: 10.1002/ejhf.1710. Epub 2019 Dec 28. PMID 31883356

RESULTS

PARTICIPANT FLOW:
Groups:
- FCM (Ferric Carboxymaltose): Ferric carboxymaltose (FCM), administered by bolus intravenous (IV) injection at a dose of 10 ml or 20 ml of undiluted solution (containing 500 mg or 1,000 mg of iron respectively) depending on the participant's body weight and haemoglobin (Hb) level.
  From a single dose given at Visit 2 (Week 0) up to 4 doses given over 24 weeks (at Visit 2 (Week 0), Visit 3 (Week 6), Visit 4 (Week 12) and Visit 5 (Week 24), depending on the participant's Hb levels measured prior to planned dosing dates.
- Placebo (Normal Saline (NaCl 0.9%)): Normal saline (NaCl 0.9%), administered by bolus intravenous (IV) injection at a volume corresponding to the FCM dose determined by the participant's body weight and haemoglobin (Hb) level (i.e., 10 ml or 20 ml per administration).
  From a single dose given at Visit 2 (Week 0) up to 4 doses given over 24 weeks (at Visit 2 (Week 0), Visit 3 (Week 6), Visit 4 (Week 12) and Visit 5 (Week 24)), depending on the participant's Hb levels measured prior to planned dosing dates.
Period: Overall Study
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Started (All Randomised Set) | 567 | 565
Started Treatment | 559 | 551
Completed | 427 | 437
Not Completed | 140 | 128
Not completed — Adverse Event | 0 | 1
Not completed — Death | 98 | 95
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 6 | 10
Not completed — Withdrawal by Subject | 27 | 15
Not completed — Other | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%)) | Total
Number analyzed (Participants) | 559 | 551 | 1110
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 64 years | 139 | 142 | 281
  Between 65 and 84 years | 369 | 370 | 739
  ≥ 85 years | 51 | 39 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 250 | 494
  Male | 315 | 301 | 616
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 50 | 101
  Not Hispanic or Latino | 498 | 489 | 987
  Unknown or Not Reported | 10 | 12 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 24 | 24 | 48
  Brazil | 14 | 14 | 28
  Croatia | 39 | 43 | 82
  Georgia | 98 | 95 | 193
  Israel | 41 | 38 | 79
  Italy | 55 | 58 | 113
  Lebanon | 16 | 16 | 32
  Netherlands | 38 | 31 | 69
  Poland | 90 | 90 | 180
  Romania | 76 | 78 | 154
  Singapore | 23 | 22 | 45
  Spain | 12 | 12 | 24
  Sweden | 4 | 1 | 5
  Ukraine | 23 | 23 | 46
  United Kingdom | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: HF Hospitalizations and CV Death
Description: HF = Heart Failure, CV = Cardiovascular.
  The composite of recurrent HF hospitalizations and CV death up to 52 weeks after randomization
  Total hospitalisations included first and recurrent events. If a participant was hospitalised for heart failure and died within 24 h from any cardiovascular event, this was counted as one event.
Time Frame: up to 52 weeks after randomization
Population: Full Analysis Set (FAS): All randomised participants for whom administration of study treatment was started and who had at least one post-baseline visit (including calls), death or hospitalisation or who withdrew from the study after but not on the randomisation date.
  The management and follow-up of patients was affected by the COVID-19 pandemic. Participants were censored in each country on the date when the first patient with COVID-19 was reported in the respective country.
Measure: Number; unit: Events
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Events
  Full Analysis Set (FAS) | 293 | 372
  Covid-19 Sensitivity Analysis | 274 | 363
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.059, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.79, 95% CI 2-sided [0.62 to 1.01]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Covid-19 Sensitivity Analysis; Test type: Other; p = 0.024, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.75, 95% CI 2-sided [0.59 to 0.96]

2. Secondary Outcome: Recurrent CV Hospitalisations and CV Death
Description: CV = Cardiovascular
  The composite of recurrent CV hospitalisations and CV death at 52 weeks after randomisation
  Total hospitalisations included first and recurrent events. If a participant was hospitalised for a cardiovascular reason and died within 24 h of admission from any cardiovascular event, this was counted as one event.
Time Frame: up to 52 weeks after randomization
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Events
  Full Analysis Set (FAS) | 370 | 451
  COVID-19 sensitivity analyses | 350 | 440
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.050, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.80, 95% CI 2-sided [0.64 to 1.0]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); COVID-19 sensitivity analyses; Test type: Other; p = 0.024, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.77, 95% CI 2-sided [0.62 to 0.97]

3. Secondary Outcome: HF Hospitalisations
Description: HF = Heart Failure
  HF hospitalisations up to 52 weeks after randomisation analysed as recurrent event.
Time Frame: up to 52 weeks after randomisation
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Events
  Full Analysis Set (FAS) | 217 | 294
  COVID-19 sensitivity analyses | 202 | 287
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.013, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.74, 95% CI 2-sided [0.58 to 0.94]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); COVID-19 sensitivity analyses; Test type: Other; p = 0.005, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.70, 95% CI 2-sided [0.55 to 0.90]

4. Secondary Outcome: CV Mortality
Description: CV = Cardiovascular
  CV mortality analysed as time to first event at 52 weeks after randomisation.
Time Frame: at 52 weeks after randomisation.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants
  Full Analysis Set (FAS) | 77 | 78
  COVID-19 sensitivity analyses | 73 | 76
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.809, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.70 to 1.32]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Covid-19 Sensitivity Analysis; Test type: Other; p = 0.687, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.68 to 1.29]

5. Secondary Outcome: Composite of HF Hospitalisations or CV Death
Description: HF = Heart Failure, CV = Cardiovascular
  Analysed as time to first event at 52 weeks after randomisation. The number of participants with at least one HF Hospitalisation or CV Death is presented below.
Time Frame: at 52 weeks after randomisation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants
  Full Analysis Set (FAS) | 181 | 209
  COVID-19 sensitivity analyses | 175 | 205
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.030, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.66 to 0.98]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Covid-19 Sensitivity Analysis; Test type: Other; p = 0.023, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.97]

6. Secondary Outcome: Days Lost Due to HF Hospitalisation or CV Death
Description: HF = Heart Failure, CV = Cardiovascular
  Number of days lost due to heart failure hospitalisations or cardiovascular death corresponds to the total number of days in hospital for heart failure from randomisation to last known date. Days lost due to cardiovascular death are added to the number of days lost due to heart failure hospitalisation.
Time Frame: at 52 weeks after randomisation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
days
  Full Analysis Set (FAS) | 3.8 (9.06) | 6.2 (14.48)
  COVID-19 sensitivity analyses | 3.5 (8.18) | 6.1 (14.42)
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.035, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.67, 95% CI 2-sided [0.47 to 0.97]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Covid-19 Sensitivity Analysis; Test type: Other; p = 0.009, Negative binomial model; Negative binomial model adjusted for baseline covariates: sex, age, HF aetiology, HF duration, and country; Annualised event rate ratio (RR) = 0.61, 95% CI 2-sided [0.42 to 0.88]

7. Other Pre Specified Outcome: HF Hospitalisations
Description: HF = Heart Failure
  Number of participants with at least one HF Hospitalisation up to 52 weeks after randomisation
Time Frame: up to 52 weeks after randomisation
Population: Full Analysis Set (FAS): All randomised participants for whom administration of study treatment was started and who had at least one post-baseline visit (including calls), death or hospitalisation or who withdrew from the study after but not on the randomisation date.
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants | 142 | 178
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.006, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.92]

8. Other Pre Specified Outcome: CV Hospitalisations
Description: CV = Cardiovascular
  Number of participants with at least one CV Hospitalisation up to 52 weeks after randomisation
Time Frame: up to 52 weeks after randomisation
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants | 181 | 220
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.009, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.63 to 0.94]

9. Other Pre Specified Outcome: All-cause Mortality
Description: Number of participants who died up to 52 weeks after randomisation
Time Frame: up to 52 weeks after randomisation
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants | 98 | 96
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.944, Regression, Cox; Cox regression adjusted for sex, age, HF aetiology, HF duration, and country at baseline; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.75 to 1.31]

10. Other Pre Specified Outcome: Change From Baseline in NYHA Functional Class
Description: NYHA = New York Heart Association
  NYHA functional class was assessed as Class I, II, III, IV or V:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients. If a participant was hospitalised at any point during any post-baseline visit and did not have any NYHA assessment for this visit, then Class IV was to be imputed for the visit.
  Class V - Imputed for participants who died.
  Lower response categories are better for score NYHA.
Time Frame: at 6, 12, 24 and 52 weeks after randomisation
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Participants
  Baseline: number analyzed (Participants) | 557 | 547
  Baseline: Class I | 14 | 8
  Baseline: Class II | 255 | 240
  Baseline: Class III | 272 | 277
  Baseline: Class IV | 16 | 22
  Baseline: Class V | 0 | 0
  Week 6: number analyzed (Participants) | 516 | 514
  Week 6: Class I | 38 | 38
  Week 6: Class II | 296 | 271
  Week 6: Class III | 151 | 151
  Week 6: Class IV | 13 | 31
  Week 6: Class V | 18 | 23
  Week 12: number analyzed (Participants) | 492 | 488
  Week 12: Class I | 39 | 40
  Week 12: Class II | 296 | 267
  Week 12: Class III | 107 | 131
  Week 12: Class IV | 14 | 18
  Week 12: Class V | 36 | 32
  Week 24: number analyzed (Participants) | 492 | 495
  Week 24: Class I | 47 | 47
  Week 24: Class II | 288 | 265
  Week 24: Class III | 88 | 100
  Week 24: Class IV | 13 | 20
  Week 24: Class V | 56 | 63
  Week 52: number analyzed (Participants) | 449 | 463
  Week 52: Class I | 48 | 53
  Week 52: Class II | 234 | 223
  Week 52: Class III | 61 | 75
  Week 52: Class IV | 7 | 17
  Week 52: Class V | 99 | 95
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Full Analysis Set (FAS); Test type: Other; p = 0.196, Generalised Estimating Equations (GEE); The following variables are included in the GEE model: treatment, visit, baseline NYHA class, sex, age, HF aetiology, HF duration, and country; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.93 to 1.39]

11. Other Pre Specified Outcome: Change From Baseline in the EQ-5D-5L Questionnaire Indexed Value
Description: EQ-5D-5L: European Quality of Life-5 Dimensions-5 Levels
  The EQ 5D questionnaire consists of a health descriptive system for participants to self-classify and rate their health status on the day of administration.
  The descriptive system includes 5 items/dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, which are coded from 1 (best state) to 5 (worst state).
Time Frame: at 6, 24 and 52 weeks after randomisation
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Change from baseline in EQ-5D-5L
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
Change from baseline in EQ-5D-5L
  Week 6: number analyzed (Participants) | 476 | 465
  Week 6 | 0.05 (0.01) | 0.03 (0.01)
  Week 24: number analyzed (Participants) | 422 | 410
  Week 24 | 0.06 (0.01) | 0.05 (0.01)
  Week 52: number analyzed (Participants) | 365 | 363
  Week 52 | 0.06 (0.01) | 0.06 (0.01)
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 6; Test type: Other; p = 0.208, Mixed-effect model of repeated measures; MMRM using unstructured covariance matrix: Change score = Baseline score + Treatment + Visit + Treatment*Visit + Baseline covariates
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 24; Test type: Other; p = 0.408, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 52; Test type: Other; p = 0.999, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]

12. Other Pre Specified Outcome: KCCQ-12 Repeated-Measures Model for Analysis of Treatment Difference
Description: KCCQ = Kansas City Cardiomyopathy Questionnaire
  The KCCQ 12 is a health-related quality of life questionnaire for Heart Failure. It is a 12 item questionnaire that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge and Quality of life. Scores are generated for each domain and scaled from 0 to 100, with 0 denoting the lowest reportable health status and 100 the highest reportable health status.
Time Frame: up to 52 weeks after randomisation
Population: as for outcome 7
Measure: Mean (Standard Error); unit: KCCQ-12 score
Arm/Group | FCM (Ferric Carboxymaltose) | Placebo (Normal Saline (NaCl 0.9%))
Number analyzed (Participants) | 558 | 550
KCCQ-12 score
  Week 2: number analyzed (Participants) | 490 | 484
  Week 2 | 18.53 (1.16) | 17.24 (1.19)
  Week 4: number analyzed (Participants) | 476 | 480
  Week 4 | 21.26 (1.18) | 18.36 (1.21)
  Week 6: number analyzed (Participants) | 475 | 461
  Week 6 | 23.49 (1.20) | 19.88 (1.23)
  Week 12: number analyzed (Participants) | 439 | 451
  Week 12 | 25.57 (1.24) | 21.88 (1.26)
  Week 24: number analyzed (Participants) | 422 | 413
  Week 24 | 26.30 (1.26) | 23.32 (1.27)
  Week 36: number analyzed (Participants) | 386 | 379
  Week 36 | 25.78 (1.28) | 23.70 (1.30)
  Week 52: number analyzed (Participants) | 368 | 370
  Week 52 | 25.75 (1.33) | 24.31 (1.34)
Statistical Analysis 1: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 2; Test type: Other; p = 0.227, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 4; Test type: Other; p = 0.018, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 6; Test type: Other; p = 0.005, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 12; Test type: Other; p = 0.006, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 24; Test type: Other; p = 0.028, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 36; Test type: Other; p = 0.136, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: FCM (Ferric Carboxymaltose) vs Placebo (Normal Saline (NaCl 0.9%)); Week 52; Test type: Other; p = 0.329, Mixed-effect model of repeated measures; [statistical method as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: During treatment period up to 52 weeks after randomization
Groups:
- Group 1 - FCM (Ferric Carboxymaltose): Ferric carboxymaltose (FCM), administered by bolus IV injection at a dose of 10 ml or 20 ml of undiluted solution (containing 500 mg or 1,000 mg of iron respectively) depending on the subject's body weight and Hb level.
  From a single dose given at Visit 2 (Week 0) up to 4 doses given over 24 weeks (at Visit 2 (Week 0), Visit 3 (Week 6), Visit 4 (Week 12) and Visit 5 (Week 24)), depending on the subject's Hb levels measured prior to planned dosing dates.
- Group 2 - Placebo (Normal Saline (NaCl 0.9%)): Normal saline (NaCl 0.9%), administered by bolus IV injection at a volume corresponding to the FCM dose determined by the subject's body weight and Hb level (i.e., 10 ml or 20 ml per administration).
Arm/Group | Group 1 - FCM (Ferric Carboxymaltose) | Group 2 - Placebo (Normal Saline (NaCl 0.9%))
All-Cause Mortality (participants affected / at risk) | 99/559 | 96/551
Serious Adverse Events (participants affected / at risk) | 250/559 | 282/551
Other Adverse Events (participants affected / at risk) | 51/559 | 45/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - FCM (Ferric Carboxymaltose) (N=559) | Group 2 - Placebo (Normal Saline (NaCl 0.9%)) (N=551)
Cardiac failure (Cardiac disorders) | 116 (163) | 127 (215)
Cardiac failure acute (Cardiac disorders) | 21 (25) | 17 (23)
Cardiac failure congestive (Cardiac disorders) | 20 (32) | 23 (35)
Atrial fibrillation (Cardiac disorders) | 10 (11) | 4 (4)
Cardiac arrest (Cardiac disorders) | 8 (8) | 11 (12)
Angina unstable (Cardiac disorders) | 5 (5) | 5 (6)
Myocardial infarction (Cardiac disorders) | 5 (5) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 5 (6) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 7 (7)
Ventricular tachycardia (Cardiac disorders) | 4 (6) | 3 (3)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 8 (8)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 5 (6)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 4 (4)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 11 (11) | 15 (16)
Sepsis (Infections and infestations) | 7 (7) | 9 (9)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2)
Cellulitis (Infections and infestations) | 4 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Shewanella algae bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Death (General disorders) | 8 (8) | 13 (13)
Sudden cardiac death (General disorders) | 5 (5) | 5 (5)
Sudden death (General disorders) | 5 (5) | 7 (7)
Multiple organ dysfunction syndrome (General disorders) | 3 (4) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (3) | 4 (6)
Asthenia (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 3 (3)
Epilepsy (Nervous system disorders) | 3 (4) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 4 (4)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 6 (6)
Renal failure (Renal and urinary disorders) | 5 (5) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (3) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Presbyoesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2)
Diabetic foot (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Corneal decompensation (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Heart rate abnormal (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - FCM (Ferric Carboxymaltose) (N=559) | Group 2 - Placebo (Normal Saline (NaCl 0.9%)) (N=551)
Cardiac failure (Cardiac disorders) | 51 (57) | 45 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02937454/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02937454/SAP_001.pdf